CLINICAL TRIAL: NCT03094416
Title: An Open-label Therapeutic Efficacy Study of Tirosint (Levothyroxine Sodium) Capsules in Thyroidectomized Patients Taking Proton Pump Inhibitors
Brief Title: Levothyroxine Sodium in Thyroidectomized Patients Taking Proton Pump Inhibitors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13US-T404
Record Dates: First submitted 2017-03-17; First posted 2017-03-29 (Actual); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Hypothyroidism;Postablative
MeSH Terms: interventions — Thyroxine; Proton Pump Inhibitors; Omeprazole; Esomeprazole; Lansoprazole; Dexlansoprazole; Pantoprazole; Rabeprazole; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- levothyroxine sodium capsules (Experimental): levothyroxine sodium capsules 88 to 250 mcg/day (depending on individual needs) for 3 months
  Interventions: Drug: levothyroxine sodium capsule; Drug: Proton pump inhibitor (PPI); Drug: Levothyroxine Sodium (LT4) Tablets

INTERVENTIONS:
Drug: levothyroxine sodium capsule — after the run-in period, patients will be switched to levothyroxine sodium capsule at the same dose used during run-in
  Other Names: Tirosint
Drug: Proton pump inhibitor (PPI) — for the whole study duration all subjects will keep taking their proton pump inhibitor medication, as per prescription and as before inclusion
  Other Names: omeprazole, esomeprazole, lansoprazole, dexlansoprazole, pantoprazole, rabeprazole
Drug: Levothyroxine Sodium (LT4) Tablets — during the run-in period, subjects will continue taking their levothyroxine sodium tablet medication as per prescription and as before inclusion

SUMMARY:
This is an open-label therapeutic efficacy study of Tirosint (levothyroxine sodium) capsules in thyroidectomized patients taking proton pump inhibitors and levothyroxine, evaluating changes in serum levels of Thyroid Stimulating Hormone (TSH) upon switch to Tirosint with respect to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent duly read, signed and dated by the subject;
2. aged ≥18 and ≤65 years;
3. history of hypothyroidism due to total thyroidectomy;
4. on stable LT4 doses for at least 6 weeks at screening (≥88 mcg daily and ≤250 mcg daily);
5. TSH at screening ≥0.3 and ≤4.0 mIU/L;
6. history of gastroesophageal reflux disease or associated gastrointestinal issues on prescription PPIs (i.e. omeprazole ≥20 mg daily, or esomeprazole ≥ 20 mg daily, or lansoprazole ≥ 15 mg daily, or pantoprazole ≥ 40 mg daily) for at least 8 weeks before screening visit and for whom chronic therapy with PPIs for the next 5 months has been prescribed;
7. for women, adequate and continuative contraceptive measures until the end of the study, if not in menopause;
8. reasonable assumption of understanding the study and willingness to take part to the study and to comply with protocol requirements.

Exclusion Criteria:

1. suspected or ascertained non-compliance with LT4 or PPI therapy;
2. subject requiring changes of levothyroxine dose;
3. use of over-the-counter (OTC) PPIs;
4. history of malabsorption or history of gastric bypass surgery, short-gut syndrome, inflammatory bowel disease and other conditions of the gastrointestinal tract that may affect drug absorption (e.g. celiac disease)3;
5. multiple co-morbidities (e.g. cardiac heart failure, active arrhythmia or history of arrhythmia, particularly atrial fibrillation, uncompensated diabetes mellitus, uncorrected adrenal insufficiency, seriously compromised hepatic, renal and/or respiratory functions);
6. neoplastic pathology, active or in remission for less than 5 years (excluding the basic thyroid pathology);
7. terminal condition;
8. parenteral or assisted enteral feeding;
9. presence of any medical condition or other circumstances which would significantly affect the safety of the subject or decrease the chance of obtaining reliable data, achieving study objectives or completing the study;
10. history of alcoholism, drug abuse or psychiatric diseases that could invalidate the informed consent or limit the subject compliance with protocol requirements;
11. pregnant (positive urine pregnancy test at screening or baseline visits) or breast-feeding subject or subject planning a pregnancy in the next months;
12. known hypersensitivity to the ingredients of the preparation involved in the study3;
13. use of forbidden concomitant medications;
14. regular consumption of soy and soy derivatives, cotton seed meals, walnuts, and dietary fibres;
15. participation in other clinical studies during the 3 months prior to screening;
16. presumption of poor reliability/cooperation;
17. any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Burman, MD, Principal Investigator — Medstar Health Research Institute
Locations (9):
- United States (9):
  - California Head and Neck Specialists, La Jolla, California
  - Coastal Metabolic Research Centre, Ventura, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - NYC Health + Hospitals/ Queens, New York, New York
  - Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - Carolina Ear Nose and Throat Clinic, Orangeburg, South Carolina
  - Virginia Commonwealth University, Richmond, Virginia
  - Stonesifer Endocrine Care & Clinical Research Inc., PS, Federal Way, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sachmechi I, Lucas KJ, Stonesifer LD, Ansley JF, Sack P, Celi FS, Scarsi C, Lanzi G, Wartofsky L, Burman KD. Efficacy of Levothyroxine Sodium Soft Gelatin Capsules in Thyroidectomized Patients Taking Proton Pump Inhibitors: An Open-Label Study. Thyroid. 2023 Dec;33(12):1414-1422. doi: 10.1089/thy.2023.0382. Epub 2023 Nov 16. PMID 37885233

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject were recuited by endocrinologists, either at hospital sites or at private practices
Pre-assignment Details: Enrolled subjects underwent a run-in period of 28-42 days, that may be extended up to 4 months, until Thyroid Stimulating Hormone (TSH) normalization, if levothyroxine sodium (LT4) dose adjustments were necessary at screening visit.
Groups:
- Tirosint Capsules: During the run-in period, subjects continued taking their levothyroxine sodium tablet medication 88 to 250 mcg/day (depending on individual needs) as per prescription and as before inclusion.
  After the run-in period, at baseline visit, subjects were switched to Tirosint (levothyroxine sodium) capsules at the same dose used during run-in and for 3 months (treatment period).
  For the whole study duration (run-in and treatment period), subjects kept taking their proton pump inhibitor medication, as per prescription and as before inclusion.
Period: Run-in
Arm/Group | Tirosint Capsules
Started | 66
Completed | 47
Not Completed | 19
Not completed — Screening failure | 8
Not completed — Sponsor Decision To Discontinue Due To Global Covid-19 Pandemic | 8
Not completed — Withdrawal by Subject | 3
Period: Treatment Period
Arm/Group | Tirosint Capsules
Started | 47
Completed | 45
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: intention to treat (ITT)
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.38 (11.111)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Peru | 1
  Black or African American | 6
  Puerto Rican | 1
  Ecuadorian | 1
  Multiracial | 1
  White | 32
  Asian | 3
  American Indian or Alaska Native | 1
  Hispanic | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47
Thyroid Stimulating Hormone (TSH) [Mean (Standard Deviation); unit: mIU/L] | 1.341 (1.5054)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI)
  kg/m^2 | 32.25 (8.286)

OUTCOME MEASURES:

1. Primary Outcome: Thyroid Stimulating Hormone (TSH)
Description: Change in Serum Levels of TSH (Thyroid Stimulating Hormone) from Baseline
Time Frame: baseline and 12 weeks
Population: intention to treat (ITT), 4 subjects not considered in the analysis because of drop-out or LT4 dose change
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 43
mIU/L | -0.676 (1.3181)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — Normal distribution of data was tested with Shapiro Wilks. Data were log transformed. A mixed model ANCOVA repeated measures model was used to test differences in means at Visit 4 vs baseline on original data. As covariates the following baseline variables were considered: Age, Sex, BMI and the prescribed Tirosint dosage (dose/Kg); p < 0.0001, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = -0.783797, Standard Error of Mean 0.158271

2. Secondary Outcome: Free Thyroxine (FT4)
Description: Change in Serum Levels of FT4 (free thyroxine) from Baseline
Time Frame: baseline and 12 weeks
Population: ITT, 4 subjects not considered in the analysis because of drop-out or LT4 dose change
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 43
pmol/L | 0.593 (2.7439)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1607, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = 0.037312, Standard Error of Mean 0.026128

3. Secondary Outcome: Total Thyroxine (TT4)
Description: Change in Serum Levels of TT4 (total thyroxine) from Baseline
Time Frame: baseline and 12 weeks
Population: ITT, 4 subjects not considered in the analysis because of drop-out or LT4 dose change
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 43
nmol/L | 2.558 (27.2426)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.4204, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = 3.397559, Standard Error of Mean 4.174962

4. Secondary Outcome: Free Triiodothyronine (FT3)
Description: Change in Serum Levels of FT3 (free triiodothyronine) from Baseline
Time Frame: baseline and 12 weeks
Population: ITT, 4 subjects not considered in the analysis because of drop-out or LT4 dose change
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 43
pmol/L | 0.263 (0.5716)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0062, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = 0.055199, Standard Error of Mean 0.019171

5. Secondary Outcome: Total Triiodothyronine (TT3)
Description: Change in Serum Levels of TT3 (total triiodothyronine) from Baseline
Time Frame: baseline and 12 weeks
Population: ITT, 4 subjects not considered in the analysis because of drop-out or LT4 dose change
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 43
nmol/L | 0.098 (0.3158)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — A mixed model ANCOVA repeated measures model was used to test differences in means at Visit 4 vs baseline on original data. As covariates the following baseline variables were considered: Age, Sex, BMI and the prescribed Tirosint dosage (dose/Kg). Normal distribution of data was tested with Shapiro Wilks. No data transformation was done; p = 0.0438, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = 0.100127, Standard Error of Mean 0.048171

6. Other Pre Specified Outcome: Creatine Phosphokinase (CPK)
Description: Change in Serum Levels of creatine phosphokinase (CPK) from Baseline
Time Frame: baseline and 12 weeks
Population: ITT, 6 subjects not considered in the analysis because of drop-out, LT4 dose change or laboratory test not performed
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 41
U/L | -35.073 (125.1454)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0254, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = -0.216479, Standard Error of Mean 0.093366

7. Other Pre Specified Outcome: Sex Hormone Binding Globulin (SHBG)
Description: Change in Serum Levels of SHBG (sex hormone binding globuline) from Baseline
Time Frame: baseline and 12 weeks
Population: ITT, 4 subjects not considered in the analysis because of drop-out or LT4 dose change
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 43
nmol/L | 0.884 (19.1861)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.7619, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = 0.011187, Standard Error of Mean 0.036679

8. Other Pre Specified Outcome: Ferritin
Description: Change in Serum Levels of ferritin from Baseline
Time Frame: baseline and 12 weeks
Population: ITT, 4 subjects not considered in the analysis because of drop-out or LT4 dose change
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 43
mcg/L | -6.442 (30.2390)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0655, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = -0.121537, Standard Error of Mean 0.064264

9. Other Pre Specified Outcome: Angiotensin Converting Enzyme (ACE)
Description: Change in Serum Levels of ACE (angiotensin converting enzyme) from Baseline
Time Frame: baseline and 12 weeks
Population: ITT, 9 subjects not considered in the analysis because of drop-out, LT4 dose change or laboratory test not performed
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 38
U/L | -0.395 (11.6237)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.5542, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = 0.031636, Standard Error of Mean 0.053033

10. Other Pre Specified Outcome: Triglycerides
Description: Change in triglycerides levels from Baseline
Time Frame: baseline and 12 weeks
Population: ITT, 7 subjects not considered in the analysis because of drop-out, LT4 dose change or laboratory test not performed
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 40
mmol/L | 0.075 (0.5419)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.6820, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = 0.019322, Standard Error of Mean 0.046827

11. Other Pre Specified Outcome: Cholesterol, Total
Description: Change in total cholesterol levels from Baseline
Time Frame: baseline and 12 weeks
Population: ITT, 7 subjects not considered in the analysis because of drop-out, LT4 dose change or laboratory test not performed
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 40
mmol/L | -0.198 (0.6685)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0468, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = -0.049243, Standard Error of Mean 0.024025

12. Other Pre Specified Outcome: Low Density Lipoprotein (LDL)-Cholesterol
Description: Change in low density lipoprotein (LDL)-cholesterol levels from baseline
Time Frame: baseline and 12 weeks
Population: ITT, 8 subjects not considered in the analysis because of drop-out, LT4 dose change or laboratory test not performed
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 39
mmol/L | -0.210 (0.5609)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.0203, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = -0.213171, Standard Error of Mean 0.088103

13. Other Pre Specified Outcome: High Density Lipoprotein (HDL)-Cholesterol
Description: Change in High Density Lipoprotein (HDL)-cholesterol levels from baseline
Time Frame: baseline and 12 weeks
Population: ITT, 7 subjects not considered in the analysis because of drop-out, LT4 dose change or laboratory test not performed
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 40
mmol/L | -0.029 (0.2460)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.4291, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = -0.030904, Standard Error of Mean 0.038699

14. Other Pre Specified Outcome: Very Low Density Lipoprotein (VLDL)-Cholesterol
Description: Change in Very Low Density Lipoprotein (VLDL)-cholesterol levels from baseline
Time Frame: baseline and 12 weeks
Population: ITT, 8 subjects not considered in the analysis because of drop-out, LT4 dose change or laboratory test not performed
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tirosint Capsules
Number analyzed (Participants) | 39
mmol/L | 0.049 (0.2338)
Statistical Analysis 1: Comparison: Tirosint Capsules; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.5967, Mixed Models Analysis — level of significance p-value < 0.05; Mean Difference (Final Values) = 0.025502, Standard Error of Mean 0.047802

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the whole study duration (from the signature of the informed consent until the end of the study and/or the follow-up planned period), an average of 18 weeks
Groups:
- Treatment Period: Tirosint Capsules: After the run-in period, at baseline visit, subjects were switched to Tirosint (levothyroxine sodium) capsules at the same dose used during run-in and for 3 months (treatment period).
  For the whole study duration (run-in and treatment period), subjects kept taking their proton pump inhibitor medication, as per prescription and as before inclusion.
- Run-in Period: LT4 Tablets: During the run-in period, subjects continued taking their levothyroxine sodium tablet medication 88 to 250 mcg/day (depending on individual needs) as per prescription and as before inclusion.
  For the whole study duration (run-in and treatment period), subjects kept taking their proton pump inhibitor medication, as per prescription and as before inclusion.
Arm/Group | Treatment Period: Tirosint Capsules | Run-in Period: LT4 Tablets
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 1/47 | 2/47
Other Adverse Events (participants affected / at risk) | 13/47 | 10/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period: Tirosint Capsules (N=47) | Run-in Period: LT4 Tablets (N=47)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period: Tirosint Capsules (N=47) | Run-in Period: LT4 Tablets (N=47)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to Covid-19 pandemic outbreak leading to discontinuation of subjects, primary endpoint was assessed on 43 subjects instead of 48 subjects (as planned in the sample size calculation). The a-posteriori study power is 91%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT03094416/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT03094416/SAP_001.pdf